CLINICAL TRIAL: NCT05139992
Title: COVID-19 Vaccine Response in People Living With Sickle Cell Disease
Brief Title: COVID-19 Vaccine Response in Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: ASH Research Collaborative (Other)
Collaborators: American Society of Hematology (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: ASH RC CTN 2021-00001
Record Dates: First submitted 2021-11-29; First posted 2021-12-01 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease; COVID-19
MeSH Terms: conditions — Anemia, Sickle Cell; COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort: Previously unvaccinated persons with sickle cell disease who are scheduled to receive their initial COVID-19 vaccine series as part of standard of care.
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — Vaccination against SARS-CoV-2 administered as part of standard of care

SUMMARY:
The purpose of this study is to assess the antibody response to COVID-19 vaccination in a cohort of patients with sickle cell disease (SCD) and to assess vaccine and SCD related complications around the time of vaccination.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a genetic disorder caused by a single base substitution of valine for a glutamine at the sixth amino acid of the gene encoding for the hemoglobin β chain. Patients with Hgb SS disease and other sickle hemoglobinopathies suffer from a variety of clinical complications related to this abnormal hemoglobin. These clinical manifestations include hemolytic anemia, painful vaso-occlusive crisis, and end organ damage. Persons with SCD generally auto-splenectomize in childhood secondary to infarctions from their hemoglobinopathy, thus increasing their risk of infection and rendering them immunosuppressed. Data suggest that general immune function in SCD patients may be impaired, and thus responses to vaccine may be suboptimal.

Patients with SCD are considered at increased risk of complications from infection from SARS-CoV-2 infection and are therefore an important group to receive vaccination against the virus. Understanding response to COVID-19 vaccination is this high-risk group of patients can provide a more targeted approach to vaccination in order to achieve adequate protection.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sickle cell disease (HbSS, HbSC, HbSB0 thalassemia, HbSB+ thalassemia, HbS/Other)
2. Has not received any COVID-19 vaccination prior to enrollment
3. Scheduled for a COVID-19 vaccination (type does not matter) as part of routine clinical care
4. Willing and able to sign consent

Exclusion Criteria:

1. Unwilling to have labs drawn or complete study requirements.
2. Previous therapy curative of SCD (including bone marrow transplant and gene therapy)
3. Previous receipt of anti-COVID-19 antibody therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 200 subjects with sickle cell disease will be enrolled at up to 20 sites participating in the ASH RC Sickle Cell Disease Clinical Trials Network.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Abrams, MD, Principal Investigator — University of Pennsylvania; Sophie Lanzkron, MD, Principal Investigator — Johns Hopkins University
Locations (8):
- United States (8):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - Montefiore Hospital, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Prisma Health - Upstate, Greenville, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anderson AR, Strouse JJ, Manwani D, Brandow AM, Vichinsky E, Campbell A, Leavey PJ, Nero A, Ibrahim IF, Field JJ, Baer A, Soto-Calderon H, Vincent L, Zhao Y, Santos JJS, Hensley SE, Mortier N, Lanzkron S, Neuberg D, Abrams CS. COVID-19 mRNA vaccination responses in individuals with sickle cell disease: an ASH RC Sickle Cell Research Network Study. Blood Adv. 2024 Sep 10;8(17):4549-4553. doi: 10.1182/bloodadvances.2024013878. PMID 38991137

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observational Cohort
Started | 59
Completed | 41
Not Completed | 18
Not completed — Withdrawal by Subject | 12
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: 41 participants completing the study
Arm/Group | Observational Cohort
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 40
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Sickle Cell Genotype [Count of Participants; unit: Participants]
  HbSS | 30
  HbS/Beta zero thalassemia | 1
  HbSC | 9
  HbS/Beta plus thalassemia | 1

OUTCOME MEASURES:

1. Primary Outcome: Antibody Response to COVID-19 Vaccine in Persons With Sickle Cell Disease
Description: IgG ELISA based antibody titer to SARS-CoV-2 spike RBD antigen
Time Frame: 2 months post initial vaccination
Measure: Median (Inter-Quartile Range); unit: units per mL
Groups:
- Observational Cohort: Previously unvaccinated persons with sickle cell disease who scheduled to receive their initial COVID-19 vaccine series as part of standard of care.
Arm/Group | Observational Cohort
Number analyzed (Participants) | 41
units per mL | 32.155 [16.9 to 65]

2. Secondary Outcome: Antibody Response to COVID-19 Vaccine in Persons With Sickle Cell Disease
Description: IgG ELISA based antibody titer to SARS-CoV-2 spike RBD antigen
Time Frame: 6 months post initial vaccination
Population: 37 participants who provided a 6-month post vaccination sample
Measure: Median (Inter-Quartile Range); unit: units per mL
Groups:
- Observational Cohort: Previously unvaccinated persons with sickle cell disease who received their initial COVID-19 vaccine series as part of standard of care.
Arm/Group | Observational Cohort
Number analyzed (Participants) | 37
units per mL | 21.43 [10.32 to 57.48]

3. Secondary Outcome: Post-Vaccination Side Effect or Sickle Cell Disease Related Complication
Description: Assessed by structured telephone interview conducted 2-3 days post-vaccination
Time Frame: 2-3 days post vaccination
Measure: Number; unit: participants
Arm/Group | Observational Cohort
Number analyzed (Participants) | 41
participants
  Participants reporting at least one side effect | 20
  Participants reporting arthralgia | 4
  Participants reporting chills | 3
  Participants reporting fever | 3
  Participants reporting headache | 5
  Participants reporting myalgia | 12
  Participants reporting Nausea | 1
  Participants reporting vaccine site redness | 3
  Participants reporting vaccine site pain | 14
  Participants reporting vaso-occlusive pain | 5

ADVERSE EVENTS:
Time Frame: 6 months
Description: Per protocol, in this observational study, only Grade II or higher adverse events associated with study participation (lab draws, questionnaire completion) were recorded.
Arm/Group | Observational Cohort
All-Cause Mortality (participants affected / at risk) | 1/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ASH Research Collaborative Clinical Trial Network Participation Agreement executed between ASH Research Collaborative (Sponsor) and participating PIs & Institutions contains disclosure language.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT05139992/Prot_SAP_000.pdf